CLINICAL TRIAL: NCT04364958
Title: The Effectiveness of a Web-based Decision Aid for Patients With Generalized Anxiety Disorder: Protocol for a Randomized Controlled Trial
Brief Title: Decision Aid for Patients With Generalized Anxiety Disorder: Protocol for a Randomized Controlled Trial
Acronym: ECA-TAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Servicio Canario de Salud (Other)
Responsible Party: Principal Investigator, Lilisbeth Perestelo-Perez, Health Services Researcher, Servicio Canario de Salud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SESCS_ECA-TAG_001
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-10

CONDITIONS: Generalized Anxiety Disorder; GAD
Keywords: Generalized Anxiety Disorder; Patient decision aids; Patient-centred care; Randomized controlled trial; Shared decision making; Web-based intervention; Primary Care
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients who agree participant and will sign the informed consent, will complete the baseline assessment. Then, those allocated to the intervention group will review the web-based PtDA (shown on the computer), with the help of a researcher if necessary, and then will fill the questionnaires assessing the outcome measures in the same web interface.
  Interventions: Other: A web based-Patient Decision Aid (PtDA) (shown on the computer)
- Control group (Active Comparator): Patients allocated to the control group will receive a web-based fact sheet (one page shown on the computer) with general information on mental health as a part of usual care, and they will also complete the same questionnaires.
  Interventions: Other: A web-based fact sheet (one page shown on the computer) with general information on mental health as a part of usual care.

INTERVENTIONS:
Other: A web based-Patient Decision Aid (PtDA) (shown on the computer) — Patient decision aids (PtDAs) are tools that assist patients in making health decisions, when there is uncertainty about treatment choice, incorporating their personal preferences and values about the available treatment options. This PtDA will include information about GAD symptoms, diagnosis, causes, and benefits and risks associated to psychological and pharmacological treatments for GAD (based on the Clinical Practice Guidelines-GAD). It will also include a values clarification exercise, in which patients will have to rate the importance attributed to the different aspects of treatments (e.g., mode of administration, benefits, risks, time to improvement, probability of relapse).
  Other Names: Intervention
  Arms: Intervention group
Other: A web-based fact sheet (one page shown on the computer) with general information on mental health as a part of usual care. — Patients in the control group will receive a fact sheet (one page) with general information on mental health as a part of usual care provided by the Canary Islands Health Service.
  Other Names: Control
  Arms: Control group

SUMMARY:
The main goal of this study is assess the effectiveness of a PtDA for patients with GAD.

DETAILED DESCRIPTION:
Background: Patients with Generalized Anxiety Disorder (GAD) have concerns and needs about their health and the health care they receive. Patient decision aids (PtDAs) are tools that assist patients in making health decisions, when there is uncertainty about treatment choice, incorporating their personal preferences and values about the available treatment options. PtDAs can improve shared decision-making (SDM) and lead to better treatment outcomes. The aim of this study is to evaluate the effectiveness of a web-based PtDA for patients with GAD in primary care.

Methods and analysis: The general study design comprises two stages: i) Development of a web-based PtDA for patients with GAD, derived from an evidence-based Clinical Practice Guideline and, ii) Assessment of the effectiveness of the PtDA employing in a randomised controlled trial (RCT) design, in primary care centres of Tenerife (Spain). This RCT will be carried out with 156 patients with GAD with a score ≥8 in the GAD-7 questionnaire, comparing the PtDA to usual care (fact sheet with general information on mental health). Patients will review the PtDA accompanied by a researcher. Post-intervention survey will be administered immediately after the intervention.

The primary outcome will be decisional conflict (immediately after intervention and 3 months after intervention).

Secondary outcomes will include knowledge about GAD and its treatment (immediately after intervention and 3 months after intervention), treatment preference (immediately after intervention), actual treatment choice (3 months after intervention), concordance between preferred and chosen (3 months after intervention) decision quality with the decision-making process (3 months after intervention), and GAD symptoms (3 months after intervention).

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years) with a diagnosis of GAD (ICD-10 or DSM-V codes: 300.02; F41.1), with a score ≥8 in the GAD-7 questionnaire, with ability to speak and read Spanish, and who accept to participate and sign the informed consent

Exclusion Criteria:

* Patients with a primary diagnosis other than GAD, a score <8 in the GAD-7, those with significant physical or mental disability that prevents from completion of study activities or those participating in other trials related with GAD treatment or education, will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Decisional conflict regarding the treatment for Generalized Anxiety Disorder, measured by the Decisional Conflict Scale (DCS) | Change from Baseline at 3 months after intervention
  DCS includes 16 items and five subscales: feeling informed, clear values about benefits or risks, support, uncertainly and effective decision. Scores are transformed to a 0-100 scale, with higher scores indicating more conflict.

SECONDARY OUTCOMES:
Decisional conflict regarding the treatment for Generalized Anxiety Disorder, measured by the Decisional Conflict Scale (DCS) | Change immediately after intervention
  CS includes 16 items and five subscales: feeling informed, clear values about benefits or risks, support, uncertainly and effective decision. Scores are transformed to a 0-100 scale, with higher scores indicating more conflict.
Knowledge about the disorder and treatment alternatives | Change immediately after intervention
  A10-item scale will be include to assess patients' knowledge of the disorder and treatments based on the contents of the PtDA.
Treatment preference | Change immediately after intervention
  Assessed with one item with four response alternatives: (pharmacological treatment, psychological treatment, combined pharmacological and psychological treatment, or unsure).
Knowledge about the disorder and treatment alternatives | Change from Baseline at 3 months after intervention
  A10-item scale will be include to assess patients' knowledge of the disorder and
Actual treatment choice | Change from Baseline at 3 months after intervention
  Assessed with one item with four response alternatives: (pharmacological treatment, psychological treatment, combined pharmacological and psychological treatment, or unsure).
Concordance between preference and choice | Change from Baseline at 3 months after intervention
  Assessed by a binary variable (concordant/non-concordant) derived from the congruence between preference and choice.
Decision quality | Change from Baseline at 3 months after intervention
  Assessed by a binary variable (yes/no) defined as a combination of adequate knowledge (≥60% of correct responses) and concordance between values and intention.
GAD symptoms | Change from Baseline at 3 months after intervention
  Assessed with the Generalized Anxiety Disorder questionnaire (GAD-7)

CONTACTS AND LOCATIONS:
Overall Officials: Lilisbeth Perestelo Perez, PhD, Principal Investigator — Servicio de Evaluacion del Servicio Canario de la Salud
Locations (1):
- Servicio de Evaluación del Servicio Canario de la Salud, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and analysed during the current study will be available from the corresponding author on reasonable request. The PtDA will be available after the end of the study on the PyDeSalud website (https://www.pydesalud.com/).
Supporting Information: CSR
Time Frame: Datasests will become available as of Nov 2020 during all the study until the estimated end date of the recruitment (January 2021) and study complete (August 2021)
Access Criteria: The PtDA will be available after the end of the study on the PyDeSalud website (https://www.pydesalud.com/).
URL: https://www.pydesalud.com/

REFERENCES:
- [Derived] Ramos Garcia V, Rivero-Santana A, Penate-Castro W, Alvarez-Perez Y, Del Mar Trujillo-Martin M, Gonzalez-Pacheco H, Santos-Alvarez A, Duarte-Diaz A, Del Cura-Gonzalez MI, Perestelo-Perez L. Effectiveness of a web-based decision aid for patients with Generalised Anxiety Disorder in Spain: a randomised controlled trial. BMJ Health Care Inform. 2025 Jul 8;32(1):e101185. doi: 10.1136/bmjhci-2024-101185. PMID 40628665
- [Derived] Perestelo-Perez L, Rivero-Santana A, Ramos-Garcia V, Alvarez-Perez Y, Duarte-Diaz A, Torres-Castano A, Trujillo-Martin MDM, Del Pino-Sedeno T, Gonzalez-Gonzalez AI, Serrano-Aguilar P. Effectiveness of a web-based decision aid for patients with generalised anxiety disorder: a protocol for a randomised controlled trial. BMJ Open. 2020 Dec 10;10(12):e039956. doi: 10.1136/bmjopen-2020-039956. PMID 33303445